CLINICAL TRIAL: NCT05796700
Title: Microwave Ablation Versus Laparoscopic Hepatectomy for 3-5cm Hepatocellular Carcinoma: a Multicentre Retrospective Study
Brief Title: Microwave Ablation Versus Laparoscopic Hepatectomy for 3-5cm Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2019-348-01
Record Dates: First submitted 2023-03-03; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-04

CONDITIONS: Overall Survival; Progression-free Survival; Cost

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave Ablation (Active Comparator): According to the shape, size and location of each patient's tumor, as well as the adjacent relationship with the surrounding organs, the individual MWA scheme was pre-established. Contrast-enhanced CT (CE-CT) or contrast-enhanced magnetic resonance imaging (CE-MRI) was used to evaluate complete ablation within 3 to 5 days after ablation. If radiography suggested incomplete ablation, supplementary ablation was performed as soon as the patient's condition permitted. A cooled-shaft MW system (KY-2000, Kangyou Medical, China) was used in the procedure.
  Interventions: Procedure: Microwave Ablation
- Laparoscopic Hepatectomy (Active Comparator): The optimal surgical procedure for each patient depends on the characteristics of the tumor. Patients were placed in French position and a laparoscopic-assisted partial hepatectomy was performed under CO2 pneumoperitoneum pressure 12-14 mmHg (1 mmHg =0.133 kPa). In most cases, a 4-well or 5-well method was used under general anesthesia.
  Interventions: Procedure: Microwave Ablation

INTERVENTIONS:
Procedure: Microwave Ablation — Microwave Ablation: A minimally invasive technique for HCC, MWA has the potential to eradicate larger HCCs with larger coagulation areas and is less affected by the heat sink effect caused by vessels around the tumor.
  Laparoscopic Hepatectomy: The technique has been widely promoted worldwide with technical progress. In patients with cirrhosis, LLR has the potential advantage of reducing the risk of postoperative liver decompensation
  Other Names: Laparoscopic Hepatectomy

SUMMARY:
As the most common subtype of liver cancer (85% ~ 90%), HCC is highly malignant; thus, one of the crucial issues in HCC management is an effective therapy for tumors at an early stage, which is vital for improving the prognosis of patients. For ≤3cm HCC, ablation has been recommended by international guidelines as a first-line or alternative treatment because of similar survival outcomes and milder liver function injury with liver resection (LR). However, the appropriate treatment options for 3-5cm HCC remain controversial. Thus, none of the international guidelines recommend ablation as a first-line treatment for 3-5cm HCC. In the past few decades, treatment for HCC has tended to be less invasive, have fewer complications, and have higher cost-effectiveness. Compared with LR, laparoscopic Hepatectomy (LH) demonstrates the advancement of minimal invasion. As another minimally invasive technique for HCC, Microwave Ablation (MWA) has the potential to eradicate larger HCCs with larger coagulation areas and is less affected by the heat sink effect caused by vessels around the tumor. Many studies have identified the potential advantages of MWA over other ablation techniques. However, to date, no clinical studies have compared the efficacy of LH and MWA therapies for 3-5cm HCC with periodic progression.

ELIGIBILITY:
Inclusion Criteria:

i) age ≥18 years ii) all patients with an initial diagnosis of 3-5cm HCC(within 3 tumors, at least one 3-5cm) by histopathology iii) Child-Pugh class A or B iv) no vascular invasion or distant metastasis v) no other malignant neoplasms within the last 5 years

Exclusion Criteria:

i) age <18 years ii) Child-Pugh class ≥B iii) vascular invasion or distant metastasis iv) with other malignant neoplasms within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1585 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | More than 3 years
  OS was defined as death related to any cause and was indexed from the date of ablation or surgery until last contact or death
Progession-free survival | More than 3 years
  DFS was defined as the time interval between first treatment and recurrence or death, whichever occurred earlier.

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with the consent of the corresponding author.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data can be shared with the consent of the corresponding author.
Access Criteria: Data can be shared with the consent of the corresponding author.

REFERENCES:
- [Derived] Wang Z, Zhang H, Meng Q, Zhang DZ, Wu SS, Hong ZX, He GB, Yang H, Xiang BD, Li X, Jiang TA, Li K, Tang Z, Huang F, Lu M, Liu C, Yu XL, Cheng ZG, Liu FY, Han ZY, Dou JP, Yu J, Liang P. A multicenter case-controlled study on laparoscopic hepatectomy versus microwave ablation as first-line therapy for 3-5 cm hepatocellular carcinoma in patients aged 60 and older. Int J Surg. 2024 Mar 1;110(3):1356-1366. doi: 10.1097/JS9.0000000000000839. PMID 38320101